CLINICAL TRIAL: NCT06956820
Title: Empowering Patients to Improve Safety in Polymedication (EmPaSafe)
Brief Title: Empowering Patients to Improve Safety in Polymedication
Acronym: EmpaSafe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: University of Ljubljana (Other); RWTH Aachen University (Other); University of Patras (Other)
Responsible Party: Principal Investigator, J.J.Swen, Professor of Clinical Pharmacy & Pharmacogenetics, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL87027.058.24
Record Dates: First submitted 2025-04-11; First posted 2025-05-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Medication Management Center — The MMC that provides patient centred information on drug-drug interactions and pharmaco-genetics affecting personal polytherapy. The MMC will show a selection of high quality publicly available information such as details on different types of medications, including their uses, side effects and instructions for use, in the language of the patient. This information is targeted at an individual patient's medication profile to inform patients to better understand and deal with their personal health information, with regard to drug therapy. Patients in the Netherlands, Slovenia and Greece also will receive their PGx profile to further personalise the MMC experience.

SUMMARY:
Rationale: In current clinical practice, polypharmacy and patient empowerment are critical yet often overlooked. Polypharmacy, the chronic use of five or more drugs, poses risks such as adverse drug reactions and decreased medication adherence, especially in elderly and multimorbid patients. Despite the interconnected nature of drug-drug and drug-gene pro inter-actions, they are considered separately. Ignoring these interactions can be hazardous, yet clinical trials to investigate them are infeasible due to fast-growing complexity, variability among patients, high costs associated with large-scale studies, and ethical and logistical chal-lenges. Consequently, there is a substantial knowledge gap in managing complex medication regimens in real-life scenarios and providing guidelines to enhance patient empowerment and drug safety. The SafePolyMed project aims to develop a patient-centred framework to define, assess and manage drug-drug, drug-gene and drug-drug-gene interactions. This framework, a web-based medication management centre, will support patients in managing their therapy-related health data, enhancing education and empowerment, and improving patient safety.

Objective: To assess the impact of the developed medication management centre on patient empowerment in polypharmacy patients, thereby improving drug safety. Secondary objec-tives are to explore if the tool is able to identify patients at risk for a drug-drug-gene interaction and lower the adverse drug event rate.

Study design: The study is a proof of concept study conducted at four institutes located in Germany, Greece, Slovenia and The Netherlands. Polypharmacy patients will use the medi-cation management centre (MMC), which provides curated, patient-specific information about drug interactions and PGx. To assess patient empowerment, patients will receive ques-tionnaires during a 12 week follow-up period.

Study population: 120 subjects with polypharmacy (defined as the chronic use of 5 or more drugs) of at least 18 years of age, with a first prescription for one of 10 index drugs. The study will be performed at 4 different sites (Leiden (NL), Patras (GR), Ljubljana (SL), Aachen (DE)) to represent different clinical settings across Europe. Each site will recruit 30 patients.

Intervention: The MMC that provides patient centred information on drug-drug interactions and pharmacogenetics affecting personal polytherapy. The MMC will show a selection of high quality publicly available information such as details on different types of medications, includ-ing their uses, side effects and instructions for use, in the language of the patient. This infor-mation is targeted at an individual patient's medication profile to inform patients to better un-derstand and deal with their personal health information, with regard to drug therapy. Patients in the Netherlands, Slovenia and Greece also will receive their PGx profile to further personal-ise the MMC experience.

Main study parameters/endpoints: The primary outcome is the sense of empowerment and health literacy for participants before and after use of the MMC. Secondary outcomes include an evaluation of the drug-drug-gene interactions and adverse drug events in the study popula-tions compared to matched historical controls.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Patients are exposed to the regular treatment. In addition, patients will receive questionnaires at baseline, two, and twelve weeks regarding the use and experience of the medication management centre, and a close-out interview at week twelve. In addition, 10ml of blood will be collected during a venipuncture for pharmacogenetic analyses.

Benefits include having access to the medication management centre for the duration of the study. Additionally, patients will receive their PGx profile. This can be used to individualize drug treatment, based on the Dutch Pharmacogenetics Working Group (DPWG) guidelines.

Overall, minimal risks are expected for subjects as they will receive normal clinical care. In-formation from the MMC will be a curation of existing publicly available data. Any information regarding DDIs and DGIs will be supplemented with a disclaimer that the patient should not adjust their treatment without talking to a healthcare provider.

ELIGIBILITY:
In order to be eligible to participate in this study, a subject must meet all of the following crite-ria:

* Polypharmacy defined as the use of 5 or more drugs
* Start usage of at least one index drug according to the list in table 3.
* Subject must be ≥ 18 years old
* Subject is able and willing to take part and be followed-up for at least 12 weeks
* Subject is able to donate blood or saliva
* Subject has signed informed consent

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactating
* Life expectancy estimated to be less than three months by treating clinical team
* Unable to consent to the study
* Unwilling to take part
* Subject has no fixed address
* Subject has previously been genotyped for PGx genes
* Subject has no current general practitioner
* Subject is, in the opinion of the Investigator, not suitable to participate in the study
* Estimated glomerular filtration rate (MDRD) of less than 15 ml/min per 1,73m2
* Patients with advanced liver failure (stage Child-Pugh C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in participants' health literacy score | 12 weeks
  Health literacy will be assessed using the Health Literacy Survey European Questionnaire (HLS-EU-Q47). Total scores range from 0 to 50, where score <26 indicates inadequate, 26-33 problematic, 34-42 adequate health literacy, and 43-50 excellent perceived health literacy. Change in total score between baseline and 12 weeks will be calculated.
  Unit of Measure: Mean change in HLS-EU-Q47 total score
Qualitative themes regarding empowerment and MMC feasibility | 12 weeks
  Semi-structured close-out interviews will be conducted to explore participants' experiences related to empowerment and health literacy after using the MMC. Interviews will be transcribed and analyzed using thematic analysis.
  Unit of Measure: Presence of major qualitative themes identified through thematic coding

SECONDARY OUTCOMES:
Accuracy of the MMC in identifying patients at risk for drug-drug-gene interactions | 12 weeks
  MMC performance will be compared to historical control data from the U-PGx cohort for identifying patients at risk for drug-drug-gene interactions.
  Unit of Measure: Sensitivity (%), specificity (%), and concordance rate (%) of MMC predictions compared to U-PGx control data
Incidence of clinically relevant adverse drug reactions (ADRs) following integration of the MMC into healthcare | 12 weeks
  The number of participants reporting one or more clinically relevant adverse drug reactions (ADRs) will be recorded and compared to matched historical controls from the U-PGx cohort.
  ADRs are defined as reactions that are:
  * causally related to the drug of inclusion (definite, probable, or possible),
  * clinically relevant (CTCAE Grade 2-5), ADRs will be identified via PRO-CTCAE responses and health complaints reported through the MMC's integrated PROMs system.
  Unit of Measure:
  Incidence rate (%) of patients reporting ≥1 clinically relevant ADR
Severity of clinically relevant adverse drug reactions (ADRs) following integration of the MMC into healthcare | 12 weeks
  Severity of ADRs will be assessed using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE).
  ADRs are defined as reactions that are:
  * causally related to the drug of inclusion (definite, probable, or possible),
  * clinically relevant (CTCAE Grade 2-5), and
  * associated with a drug-genotype interaction (as per DPWG guidelines).
  * PRO-CTCAE responses are rated on a 0-4 Likert scale, with higher scores indicating greater severity.
  Unit of Measure:
  Mean PRO-CTCAE severity score (scale 0-4; higher = more severe)

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (2):
  - Universitatsklinikum Aachen, Aachen
  - Universitatsklinikum Heidelberg, Heidelberg
- University Hospital Patras, Pátrai, Greece
- University Hospital Ljubljana, Ljubjana, Slovenia

DOCUMENTS (1):
  • Study Protocol (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/20/NCT06956820/Prot_000.pdf